CLINICAL TRIAL: NCT03985124
Title: A Randomized Controlled Trial of Tuning in to Kids in Norwegian FUS Kindergartens
Brief Title: Tuning in to Kids in Norwegian FUS Kindergartens
Acronym: TIK-FUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Sophie Havighurst, Associate Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2019-03-19; First posted 2019-06-13 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Emotional Intelligence

STUDY DESIGN:
Intervention Model Description: Cluster randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention TIK-T (Experimental): 24 kindergartens will receive the full intervention. Dosage: 1 3 hour implementation session for kindergarten leaders; 1 x 2-day training workshop for kindergarten leaders and a lead resource person in each kindergarten who will support teachers in learning and implementing Emotion Coaching with children; 2 full training days for all teachers/childcare workers in Emotion Coaching; 2 x booster sessions for all teachers with the resource person in their kindergarten to assist them in using Emotion Coaching with children in their kindergartens.
  Interventions: Behavioral: Tuning in to Kids for Teachers
- wait list control (No Intervention): 24 kindergartens will be in the 12-month wait list condition

INTERVENTIONS:
Behavioral: Tuning in to Kids for Teachers — This is an emotion-focused intervention for teachers giving them skills in emotion coaching children in their care and also understanding and managing their own emotions.
  Arms: Intervention TIK-T

SUMMARY:
The proposed project will aim to evaluate the impact of the Tuning in to Kids program for teachers using a randomised controlled research design with 48 kindergartens across Norway (Oslo, Trondheim and Bergen). Kindergartens will be randomised into intervention or 12-month wait list control. Measures will be given to kindergarten leaders, teachers, parents and in a subset of kindergartens children. Intervention kindergartens will receive training in how to be more emotion coaching as well as helping teachers understand and manage their own emotions. Primary outcomes are teachers' responsiveness to children's emotions and the overall classroom functioning/climate. Secondary outcomes are impacts on kindergarten functioning, staff absences/turn over, parents reports of children's emotional, behavioural and social functioning.

DETAILED DESCRIPTION:
The research questions will be does Tuning in to Kids (TIK) for teachers:

1. lead to improved teacher meta-emotion philosophy (beliefs about emotions), teacher emotion awareness/regulation and wellbeing?
2. lead to improved teacher emotion socialisation (decreased emotion dismissiveness and increased emotion coaching) and emotional responsiveness?
3. lead to improvements in the kindergarten social and emotional climate and improved organisational functioning of the kindergarten?
4. lead to improved child emotion vocabulary and social, emotional, behavioural functioning?
5. provide a cost-effective method for improving the functioning of the FUS kindergartens?

TIK for Teachers will aim to alter the teacher and kindergarten functioning which in turn is expected to impact children's emotional competence (emotion vocabulary/regulation) thereby impacting wider aspects of child functioning (behaviour, social functioning). In this trial of Tuning in to Kids in Norwegian FUS kindergartens, a cluster randomised design will be used. Forty-eight kindergartens, (consisting of 880 teachers), will be randomised into intervention or 12-month wait-list control. All kindergartens (intervention and control) will complete measures at baseline and 10-month follow-up (in August 2019 and then June 2020). Once baseline measures have been collected from all kindergartens (intervention and control), those in the intervention condition will receive the TIK intervention (October through to March). Twelve-month follow up measures will be collected in June 2020 and will be the same measures collected at baseline (outlined below) as well as data on intervention implementation (attendance dosage, feasibility, acceptability). Control kindergartens will receive the same measures at the same times as the intervention kindergartens and will receive the intervention after the 12-month waiting period (in autumn 2020).

Tuning in to Kids for Teachers - TIK-T: Intervention

This intervention is professional training for teachers/childcare workers. Key components include:

* Kindergarten leaders/principals and all school workers will receive an initial three hour briefing on the intervention in March 2019;
* Kindergarten leaders/lead pedagogue will attend a two-day (14 hours) professional training in TIK to learn to use emotion coaching with children in December 2019. This will give them skills to support teachers in their application of the ideas in their interactions with children.
* Childcare workers/kindergarten teachers will attend a full day training (seven hours) in how to use emotion coaching and in skills to understand and regulate their emotions January 2020;
* The Kindergarten leaders/education or pedagogue will deliver supervision sessions to assist teachers in implementation of the TIK ideas. This will be two x three hour sessions at monthly intervals (February, March 2020);
* Structured manuals will be used for intervention delivery and fidelity checklists to ensure adherence to the intervention.
* Support materials will be provided in online format/manuals for all teachers.

Measures:

* a structured, validated observation measure of classroom social-emotional environment;
* teacher responses on questionnaires about their meta-emotion philosophy (beliefs about emotions), emotion awareness/regulation, emotion socialisation (emotion dismissiveness and emotion coaching), emotion wellbeing/mental health and perceptions of the functioning of the kindergarten/school;
* kindergarten leader's responses on questionnaires about the kindergarten environment;
* kindergarten organisational data on teacher absences, staff turnover etc to measure overall organisational functioning;
* parents will complete an online questionnaire about their child's emotional language, social/emotional/behavioural functioning and their experience of support/engagement with the kindergarten. The will also complete a brief measure on their emotion socialization.
* a small number of children (for whom parental consent is given) in eight kindergartens will participate in a direct assessment at the kindergarten of the child's emotion knowledge;
* costs of intervention delivery along with expected financial costs/benefits of (improved) organisational functioning (such as costs of staff absences, re-hiring, organisational problems)
* Intervention implementation: information will be collected from teachers/kindergarten leaders about intervention acceptability, feasibility and dosage/attendance.

ELIGIBILITY:
Inclusion Criteria:

* teachers/kindergarten workers in the eligible kindergartens
* all children

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1300 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Change in Coping with Toddler's Negative Emotions Scale (CTNES) | Baseline and 10 month follow up
  Teacher's responsiveness to children's emotions using the CTNES (12 scenarios, 6 possible responses for each)
Change in Classroom Assessment Scoring System (CLASS) | Baseline and 10 month follow up
  The CLASS" is an observational tool for assessing classroom quality in the kindergarten based on teacher - child interactions in the classroom rather than evaluation of the physical environment or a specific curriculum. Divided into 3 domains: emotional support (positive climate, negative climate, teacher sensitivity, and regard for student perspectives), classroom organization (behavior management, productivity, and instructional learning formats), and instructional support (concept development, quality of feedback, and language modeling). These constructs are rated on a 7-point scale (1-2 low, 3-5 mid, and 6-7 high) recorded in 30-minutes (20 min observation, 10 min scoring) cycles over a period of up to 3 hours (with six as the recommended average number of observation cycles).

SECONDARY OUTCOMES:
Change on Brief Problem Monitor (BPM) | Baseline and 10 month follow up
  Parent reports on children's behavioural functioning using the BPM, an 18-item parent-reported questionnaire. Items are rated on a 0, 1, 0r 2 scale, with one being absence and 2 being strongly indicated.
Change on Emotion Regulation Checklist, | Baseline and 10 month follow up
  Parent report on child emotion regulation; a 24 item parent reported questionnaire that gives subscales of emotion regulation and lability/negativity.
Change on EAS Temperament Scale | Baseline and 10 month follow up
  Parent report on child emotionality using a 20 item measure that gives subscales of Reactivity, Sociability, Shyness and Activity
Change on Emotional literacy - parent reported | Baseline and 10 month follow up
  Parent report emotion language using a list of 60 emotion words where parents indicate whether or not the child would understand the given word.
Change on Emotional literacy - direct assessment | Baseline and 10 month follow up
  Using an iPad, and 60 different emotion words, testers will ask the child to point to one of 4 pictures to see if they can identify emotion words.
Change on Parent perception of kindergarten environment | Baseline and 10 month follow up
  Questions about perceived emotional support child receives in kindergarten. These will be set questions asking parents to rate on a 1 - 5 point likert scale their satisfaction, support etc from the kindergarten.
Change on Teacher perception of kindergarten environment | Baseline and 10 month follow up
  Questions about perceived support teacher received in workplace. These will be set questions asking teachers to rate on a 1 - 5 point likert scale their satisfaction, support perceived functioning of the kindergarten.

CONTACTS AND LOCATIONS:
Overall Officials: Evalill B Karevold, PhD, Study Chair — University of Oslo
Locations (3):
- Norway (3):
  - FUS Kindergartens, Bergen
  - FUS Kindergartens, Oslo
  - FUS Kindergartens, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skaland VR, Havighurst SS, Nygaard E, Teig IL. Qualitative evaluation of the implementation of "Tuning in to Kids" in Norwegian Kindergartens. BMC Psychol. 2023 Mar 30;11(1):87. doi: 10.1186/s40359-023-01088-4. PMID 36998061